CLINICAL TRIAL: NCT01722019
Title: Prospective Multicentric Randomised Trial Between Radiofrequency Ablation With VNUS Closure Fast ® and Endovenous Ablation With 1470 nm Diod Laser and Tulip Fiber ® for Treatment of Primary Venous Insufficiency.
Brief Title: Prospective Multicentric Trial Between Radiofrequency Ablation With VNUS Closure Fast ® and Endovenous Ablation With 1470 nm Diode Laser and Tulip Fiber ® for Treatment of Primary Venous Insufficiency.
Acronym: VNUS vs TULIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: European Venous Forum. (Unknown); Benelux Society of Phlebology. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/693
Record Dates: First submitted 2012-10-29; First posted 2012-11-06 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Chronic Venous Insufficiency C2 or Higher
Keywords: venous insufficiency
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- radiofrequency ablation with VNUS closure fast (Active Comparator): Radiofrequency ablation will be performed with VNUS closure fast.
  Interventions: Device: VNUS closure fast
- laser ablation and Tulip fiber (Experimental): Laser ablation with a 1470 nm wave length in combination with a new fiber, the Tulip fiber.
  Interventions: Device: Tulip fiber

INTERVENTIONS:
Device: Tulip fiber — Laser ablation with a wavelength of 1470 nanometers will be performed, in combination with a new sort of fiber: the tulip tip fiber.
  Arms: laser ablation and Tulip fiber
Device: VNUS closure fast — Radiofrequent ablation will be performed in combination with the catheter 'VNUS closure fast'.
  Arms: radiofrequency ablation with VNUS closure fast

SUMMARY:
Endovenous ablation of the greater saphenous vein has nowadays the same outcome as open crossectomy and stripping. The two most performed techniques for endovenous ablation are the endovenous laser ablation and the radiofrequency ablation. According to the trial of Rasmussen, they are equivalent for occlusion but the lower laser wave lengths resulted in more pain and paresthesia. The newer wave length of 1470 nm showed lesser side effects in observational studies. The aim of this study is to compare radiofrequency ablation with the VNUS closure fast ® with laser ablation with a 1470 nm wave length in combination with a new fiber, the Tulip fiber ®. This fiber has the shape of a tulip at his tip which avoids point necroses of the vessel wall and on consequence results in lesser side effects from wall perforations such as pain, haematoma,…

ELIGIBILITY:
Inclusion Criteria:

* Endovenous ablation of the great saphenous vein (GSV) planned
* Patient signed informed consent
* Patient must complete the 1 year follow-up
* CEAP between 2 and 6
* BMI=<35
* Diameter of the GSV in upward position less than 20 mm diameter
* No problems in deep venous system

Exclusion Criteria:

* No informed consent is signed
* Latex allergy
* Arterial insufficiency
* Deep vein thrombosis or deep vein insufficiency
* Klippel Trenaunay
* Diameter fo GSV > 20 mm
* Cross dilation with 2 or more insufficient side branches
* Previous GSV operation
* Redo-operation
* Carcinoma less than 1 year ago
* BMI > 35
* Liver-insufficiency with contraindication for local tumescence
* Intake of warfarins
* Pregnancy, breastfeeding, < 3 months after pregnancy
* Bilateral GSV insufficiency that has to be treated
* Cross insufficiency of the accessory saphenous vein or insufficiency of the subterminal valve of the GSV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Closure of the greater saphenous vein at 12 months. | 12 months after procedure
  Closure of the greater saphenous vein will be measured by venous duplex, Kabnick score and modified Gelev score. This will be performed after 5 days, 1 month, 6 months and 12 months.

SECONDARY OUTCOMES:
Pain. | after 5 days
  This will be measured with the VAS score, VCSS score, CIVIQ score, clinical evaluation and hematoma score.
Pain. | after 14 days
  This will be measured with the VAS score, VCSS score, CIVIQ score, clinical evaluation and hematoma score.
Pain. | after 1 month
  This will be measured with the VAS score, VCSS score, CIVIQ score, clinical evaluation and hematoma score.
Pain. | after 6 months
  This will be measured with the VAS score, VCSS score, CIVIQ score, clinical evaluation and hematoma score.
Pain. | after 1 year.
  This will be measured with the VAS score, VCSS score, CIVIQ score, clinical evaluation and hematoma score.
Patient satisfaction rate. | after 5 days
  This will be measured with the VAS score, VCSS score, CIVIQ score, clinical evaluation and hematoma score.
Patient satisfaction rate. | After 14 days.
  This will be measured with the VAS score, VCSS score, CIVIQ score, clinical evaluation and hematoma score.
Patient satisfaction rate. | After 1 month
  This will be measured with the VAS score, VCSS score, CIVIQ score, clinical evaluation and hematoma score.
Pain satisfaction rate. | After 6 months
  This will be measured with the VAS score, VCSS score, CIVIQ score, clinical evaluation and hematoma score.
Patient satisfaction rate. | After 1 year.
  This will be measured with the VAS score, VCSS score, CIVIQ score, clinical evaluation and hematoma score.
Incapacity to work. | after 5 days
  This will be measured with the VAS score, VCSS score, CIVIQ score, clinical evaluation and hematoma score.
Incapacity to work. | After 14 days
  This will be measured with the VAS score, VCSS score, CIVIQ score, clinical evaluation and hematoma score.
Incapacity to work. | After 1 month
  This will be measured with the VAS score, VCSS score, CIVIQ score, clinical evaluation and hematoma score.
Incapacity to work. | After 6 months
  This will be measured with the VAS score, VCSS score, CIVIQ score, clinical evaluation and hematoma score.
Incapacity to work. | After 1 year
  This will be measured with the VAS score, VCSS score, CIVIQ score, clinical evaluation and hematoma score.

CONTACTS AND LOCATIONS:
Overall Officials: Carend Randon, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (3):
- Belgium (3):
  - Ghent University Hospital, Ghent
  - University Hospital Leuven, Leuven
  - Sint-Andriesziekenhuis Tielt, Tielt

REFERENCES:
- See also: Related Info — http://www.uzgent.be